CLINICAL TRIAL: NCT04035876
Title: A Single Group, Open Label, Multi-center Clinical Study of Combination Camrelizumab (SHR-1210) and Apatinib for Downstaging/Bridging of Hepatocellular Cancer Before Liver Transplant
Brief Title: Combination Camrelizumab (SHR-1210) and Apatinib for Downstaging/Bridging of HCC Before Liver Transplant
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Shulan (Hangzhou) Hospital (Other); West China Hospital (Other); Huashan Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); The First Hospital of Jilin University (Other); Tianjin First Central Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiao Xu, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2019-SHR-APA-ZJU
Record Dates: First submitted 2019-07-20; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Hepatocellular Carcinoma; Liver Transplant
Keywords: Camrelizumab; Apatinib; HCC; Liver transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab plus apatinib (Experimental)
  Interventions: Drug: Camrelizumab plus apatinib

INTERVENTIONS:
Drug: Camrelizumab plus apatinib — Camrelizumab 200mg q2w iv and apatinib 250mg qd po.

SUMMARY:
To assess the primary effects and safety of camrelizumab (SHR-1210) plus apatinib for downstaging/bridging of HCC before liver transplantation.

DETAILED DESCRIPTION:
HCC patients waiting for liver transplantation will be screened and enrolled according to the inclusion criteria. After screening and enrollment, patients will be administrated camrelizumab 200mg q2w iv and apatinib 250mg qd po regimen every 4 weeks as a cycle. Each patient will receive camrelizumab treatment for at least 2 cycles and discontinue camrelizumab 5 weeks before liver transplantation. Apatinib will be discontinued 1 week before liver transplantation. Once the tumor progression was detected, the program will be terminated and the appropriate optimal treatment will be given. The objective remission rate (ORR), recurrence-free survival (RFS), overall survival (OS), time to progress (TTP) and any adverse effect during the study will be evaluated in order to assess the primary effects and safety of camrelizumab (SHR-1210) plus apatinib for downstaging/bridging of HCC before liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* Pathology: hepatocellular carcinoma
* Exceed Hangzhou Criteria (Type A: diameter of tumor ≤ 8 cm or diameter of tumor and AFP ≤ 100 ng/mL; Type B: diameter of tumor >8 cm, but 100 ng/mL < AFP <400 ng/mL)
* No interventional therapy (TACE, RFA or I131) within 2 month
* Expected survival for more than 3 months
* Child-pugh grade A or grade B (≤ 7 points)
* Absolute neutrophil count ≥ 1.5×10^9 /L, Hb ≥ 9 g/L, PLT ≥ 100×10^9 /L; TSH ≤ ULN; total bilirubin ≤ 1.5 ULN, albumin ≥ 28 g/L, AST, ALT ≤ 3 ULN; serum creatinine ≤ 1.5 ULN
* ECOG: 0-2
* Patients participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Regional lymph node metastases or extrahepatic metastases
* Allergic to Camrelizumab or Apatinib
* Patients who have had or are currently complicated with other malignant tumors
* Active hepatitis (hepatitis B: HBsAg positive or HBV- DNA≥10⁴copies/ml; hepatitis C: HCV antibodies and HCV-RNA positive)
* Activ pulmonary tuberculosis or pulmonary tuberculosis history
* Active, diagnosed, or suspected autoimmune disease (including but not limited to: uveitis, enteritis, hepatitis, pituitary, nephritis, vasculitis, hyperthyroidism, hypothyroidism and asthma)
* Interstitial lung disease history or non-infectious pneumonia requiring oral or intravenous steroid therapy
* Long-term systemic hormone therapy (dose > 10mg prednisone/day) or any other form of immunosuppressive therapy
* Myocardial ischemia or myocardial infarction above grade II, hypertension and inability to reach the normal range after medication (systolic blood pressure >140mmHg, diastolic blood pressure >90mmHg)
* Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg<2g/L); history of gastrointestinal bleeding within 6 months; obvious bleeding tendency or undergoing thrombolytic or anticoagulant treatment
* Pregnant or lactating women
* Patients who participated in other clinical trials within 1 month
* Active infections which require systemic treatment
* HIV positive
* Other factors that may affect patients' safety or compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-16 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate | From enrollment to disease progression, up to 6 months
  The proportion of patients with CR, PR, and SD in the group
Recurrence-free survival | 1 year
  The period from enrollment surgery to recurrence of HCC

SECONDARY OUTCOMES:
Overall survival | 1 year
  The survival rate in a year
Time to progress | From enrollment to disease progression, up to 6 months
  The period from enrollment to disease progression
Adverse effect | 1 year
  Any adverse effects occur during the project

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No